CLINICAL TRIAL: NCT02019329
Title: A SINGLE-CENTER, RANDOMIZED, INVESTIGATOR/SUBJECT-BLIND, MULTIPLE-DOSE, PLACEBO-CONTROLLED, PARALLEL STUDY TO INVESTIGATE THE SAFETY, TOLERABILITY AND PHARMACOKINETICS OF RO5545965 IN PATIENTS WITH SCHIZOPHRENIA ON RISPERIDONE.
Brief Title: A Study of the Safety, Tolerability and Pharmacokientics of RO5545965 in Patients With Schizophrenia on Risperidone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP29188
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo + risperidone (Placebo Comparator)
  Interventions: Other: Placebo; Drug: risperidone
- RO5545965 + risperidone (Experimental)
  Interventions: Drug: RO5545965; Drug: risperidone

INTERVENTIONS:
Other: Placebo — Oral daily administration from Days 1-12
  Arms: Placebo + risperidone
Drug: RO5545965 — Oral daily administration from Days 1-12
  Arms: RO5545965 + risperidone
Drug: risperidone — 13 day run-in phase until 4 mg daily dose level is reached. 4 mg daily oral dose until Day 17 of study, for a total of 30 days. Dose may be increased up to 6 mg at the investigator's discretion. After study treatment, risperidone dosage may be decreased, increased or omitted at the investigator's discretion during a wash-out phase while patients return to their chronic antipsychotic treatment. Patient response during wash-out will be monitored in-house for 48 hours after the last dose of RO5545965 or placebo is administered. This in-house observation may be extended as needed by the investigator.

SUMMARY:
This randomized, double-blinded, placebo-controlled study will investigate the safety, tolerability, and pharmacokinetics of multiple doses of RO5545965 administered orally to psychiatrically stable patients with schizophrenia receiving risperidone.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged >/= 18 years and </= 60 years
* Clinically stable, mild or moderate schizophrenia
* On stable antipsychotic treatment for the last 6 months
* Generally healthy in the investigator's opinion, based on assessment of medical history, physical examination, vital signs, electrocardiogram (ECG), and the results of the hematology, clinical chemistry, urinalysis, serology, and other laboratory tests
* Willingness to be hospitalized for approximately 3 weeks
* BMI > 18.5 kg/m2 and < 38 kg/m2
* Use of highly effective contraception as defined by the study protocol. Men must also not donate sperm until at least 30 days after the last dose, and women cannot be pregnant or breastfeeding

Exclusion Criteria:

* Treatment with antiparkinson medication including anticholinergic drugs
* Treatment with depot antipsychotic medication within the last three months prior to screening
* Participation in a clinical trial with an investigational drug or device < 3 months prior to screening
* Smokes more than 20 cigarettes per day
* Current drug abuse (excluding nicotine) or drug abuse within 3 months prior to the screening visit
* Any donation of blood or significant blood loss within three months prior to first administration of the study drug
* Use of prohibited medications (including vitamins or herbal remedies) taken within 14 days or within 5 times the elimination half-life of the medication (whichever is longer) before the first study drug administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 10 weeks
Health of the patients, assessed through a complete medical examination including physical examination, electrocardiogram (ECG) and vital signs. | Up to 10 weeks

SECONDARY OUTCOMES:
Pharmacokinetics: Plasma area under the concentration-time curve (AUC) of RO5545965 | 17 days
Pharmacokinetics: Plasma area under the concentration-time curve (AUC) of risperidone | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Glendale, California, United States